CLINICAL TRIAL: NCT05953597
Title: Effectiveness of a Nutrition Education Program in Improving Nutrition Knowledge and Related Biomarkers in Individuals with Spinal Cord Injury
Brief Title: Nutrition Education Program in Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Elizabeth Felix, Research Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20230569
Record Dates: First submitted 2023-07-10; First posted 2023-07-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries
Keywords: Metabolic dysfunction; Nutrition education
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition Education Group (Experimental): Participants in this study arm will receive nutrition education once a month for 12 months.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Nutrition Education — The intervention will consist of 12 monthly nutrition education sessions catered to people with spinal cord injuries. The curriculum is based on the 2020-2025 Dietary Guidelines for Americans such as consuming recommended amounts of fruits/vegetables, whole grains, etc. The sessions will be approximately 30-60 minutes and will be available in-person.

SUMMARY:
The purpose of this research is to assess the effectiveness of a nutrition education program in increasing nutrition knowledge and improving health-related biomarkers in individuals with spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

- Adults with SCI with complete and incomplete (American Spinal Injury Association Impairment Scale Score A-D) paraplegia or ventilator-independent tetraplegia.

Exclusion Criteria:

* Participants who do not meet inclusion criteria.
* Adults unable to consent.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women (self-report)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition Knowledge | Baseline, 12 months
  The General Nutrition Knowledge Questionnaire is an 88-item scale that has a scoring range of 0 to 88 with a high score indicating more knowledge of nutrition.

SECONDARY OUTCOMES:
Change in Cardiometabolic Biomarkers - Fasting Sodium | Baseline, 12 months
  Measured in millimoles/liter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Potassium | Baseline, 12 months
  Measured in millimoles/liter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Chloride | Baseline, 12 months
  Measured in millimoles/liter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Blood Urea Nitrogen | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Glucose | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers -Triglycerides | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Total Cholesterol | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Low Density Lipoprotein Cholesterol | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Very-low-density lipoprotein | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers -High-density lipoprotein cholesterol | Baseline, 12 months
  Measured in milligrams/deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Hemoglobin a1c | Baseline, 12 months
  Measured as a percentage of hemoglobin a1c, assessed with blood analyses.
Change in Cardiometabolic Biomarkers - Insulin | Baseline, 12 months
  Measured in units of insulin per millimeter (uU/ml) assessed with blood analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Felix, PhD, Principal Investigator — University of Miami
Locations (1):
- Christine E. Lynn Rehabilitation Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sneij A, Farkas GJ, Carino Mason MR, Gater DR. Nutrition Education to Reduce Metabolic Dysfunction for Spinal Cord Injury: A Module-Based Nutrition Education Guide for Healthcare Providers and Consumers. J Pers Med. 2022 Dec 7;12(12):2029. doi: 10.3390/jpm12122029. PMID 36556250